CLINICAL TRIAL: NCT06938516
Title: IMPACT of Nebilet in Blood Pressure Control in Patients With HYpertension: An Observational, Longitudinal Study
Brief Title: Prospective Observational Study On The Impact Of Nebilet In Blood Pressure Control In Hypertensive Patients (HYIMPACT)
Acronym: HYIMPACT
Status: Recruiting | Type: Observational
Sponsor: A.Menarini Asia-Pacific Holdings Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AMAP/22/NebHyp/001
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Nebivolol in high blood pressure; Use of Nebilet in high blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The HYIMPACT study (IMPACT of Nebilet® in Blood Pressure Control in Patients with Hypertension) is a multinational, multicenter, observational, prospective, longitudinal real-world evidence study designed to assess the effectiveness and safety of Nebilet® (nebivolol) in hypertensive patients. The study aims to evaluate changes in systolic and diastolic blood pressure from baseline to 12, 24, and 36 months, as well as treatment adherence, quality of life, prescription patterns, and cardiovascular outcomes.

A total of approximately 5,000 hypertensive patients with or without cardiovascular comorbidities will be enrolled across seven Asian countries (Malaysia, Indonesia, the Philippines, Korea, Vietnam, Thailand, and Taiwan). Patients newly initiated on Nebilet®-based treatment or already receiving Nebilet® for no more than two weeks prior to screening will be eligible for inclusion.

Patients will be followed at regular intervals for up to three years. The study will also assess the correlation between home and office blood pressure measurements and compare Nebilet® monotherapy with combination therapy in achieving target blood pressure control. The findings from this study will provide real-world insights into the clinical management of hypertension with Nebilet® and its impact on patient outcomes.

DETAILED DESCRIPTION:
Introduction. Hypertension remains one of the leading risk factors for cardiovascular morbidity and mortality worldwide, contributing significantly to the burden of stroke, heart failure, and other cardiovascular diseases. Despite advancements in antihypertensive therapies, real-world data on long-term blood pressure control, treatment adherence, and patient-reported outcomes remain insufficient, particularly in diverse populations across Asia. While clinical trials have established the efficacy of various antihypertensive agents, the applicability of these findings to routine clinical practice remains unclear. Beta-blockers, particularly nebivolol, a third-generation β1-selective adrenergic antagonist with nitric oxide-mediated vasodilatory properties, have demonstrated favorable hemodynamic effects, improved vascular function, and better tolerability compared to traditional beta-blockers. However, there is a lack of robust real-world evidence assessing its long-term impact on blood pressure control and cardiovascular outcomes.

The HYIMPACT study is a multinational, multicenter, observational, longitudinal study designed to evaluate the real-world effectiveness, safety, and adherence of Nebilet® (nebivolol) in hypertensive patients across seven Asian countries. This study will provide insights into the clinical utility of Nebilet® in achieving sustained blood pressure control over time, while also assessing the influence of cardiovascular risk factors on treatment outcomes. By systematically collecting data from patients in routine clinical settings, HYIMPACT aims to bridge the gap between controlled clinical trials and real-world practice, offering valuable evidence to optimize hypertension management strategies.

Study Objectives. HYIMPACT aims to assess the impact of Nebilet®-based treatment on systolic and diastolic blood pressure control from baseline to 12, 24, and 36 months. The study will determine the proportion of patients achieving target blood pressure levels (<140/90 mmHg) and evaluate adherence using the Morisky 8-Item Medication Adherence Scale (MMAS). Additionally, the study will compare the effectiveness of Nebilet® monotherapy versus combination therapy in achieving blood pressure control. Patient-reported outcomes will be analyzed using the SF-36 and MINICHAL questionnaires, providing insights into the impact of treatment on quality of life. The study will also assess the correlation between home and office blood pressure measurements and investigate the association between Nebilet® use and major adverse cardiovascular events (MACE), including myocardial infarction, stroke, and cardiovascular mortality.

Study Design and Population. HYIMPACT is an observational, prospective, longitudinal study enrolling approximately 5,000 hypertensive patients across Malaysia, Indonesia, the Philippines, Korea, Vietnam, Thailand, and Taiwan. Eligible patients will be adults aged 18 years or older with newly diagnosed or uncontrolled hypertension, defined as an office systolic blood pressure of at least 140 mmHg and/or diastolic blood pressure of at least 90 mmHg at screening. Patients may be included if they have either been newly prescribed Nebilet® or have been on Nebilet®-based treatment for no more than two weeks prior to enrollment. Individuals with recent major cardiovascular events within the last three months, severe heart failure classified as NYHA Class IV, or contraindications to Nebilet® as per the Summary of Product Characteristics will be excluded. The study will involve 300 to 500 physicians, ensuring representation across a wide range of real-world clinical settings.

Variables to be Collected. The study will systematically collect patient demographic and clinical data, including medical history, cardiovascular risk factors such as diabetes, obesity, and hypercholesterolemia, and medication use. Blood pressure measurements will be recorded at baseline and at each follow-up visit, with additional data collected on prescription patterns, dose adjustments, and patient adherence. Laboratory parameters, including lipid profiles, glycated hemoglobin (HbA1c), and renal function markers, will be documented when available. Cardiovascular outcomes such as MACE, including myocardial infarction, stroke, and cardiovascular mortality, will be monitored throughout the study.

Follow-Up and Data Collection. Patients will be evaluated at baseline and followed up at 12, 24, and 36 months. Blood pressure will be measured at each visit using standardized protocols, and home blood pressure readings will be encouraged to assess their correlation with office measurements. Patient-reported quality of life and adherence assessments will be conducted using validated questionnaires. Any adverse events, including treatment-emergent and serious adverse events, will be documented. Data will be recorded in an electronic case report form (eCRF) using the CLINYTICS platform, ensuring consistency and standardization across study sites.

Quality Control Measures. To ensure high data quality, the study will implement standardized definitions and data collection procedures across all sites. Investigators will receive training on study protocols, and automated validation checks within the eCRF system will help identify inconsistencies. Regular site audits will be conducted to monitor compliance, and periodic investigator meetings will be held to review study progress. Ethics committee approvals will be obtained in each participating country, and all data will be handled in compliance with Good Clinical Practice (GCP) guidelines and local data protection regulations.

Statistical Analysis. Continuous variables such as blood pressure values will be summarized as means with standard deviations, while categorical variables will be presented as frequencies and percentages. Changes in systolic and diastolic blood pressure over time will be analyzed using paired t-tests and repeated measures ANOVA, with non-parametric alternatives applied when normality assumptions are not met. The effectiveness of Nebilet® monotherapy versus combination therapy will be assessed using logistic regression for categorical outcomes and ANOVA for continuous variables. Cox proportional hazards models will evaluate the association between Nebilet® treatment and cardiovascular outcomes. Pearson correlation coefficients will be used to analyze the relationship between home and office blood pressure measurements, and structural equation modelling (SEM) will be applied to address potential regression dilution bias.

Study Governance and Data Ownership. HYIMPACT is an investigator-led study with data collection coordinated through a centralized electronic data management system. Each participating physician retains ownership of individual patient data, while consolidated and anonymized study results will be used for scientific analysis and publication. Patient confidentiality will be strictly maintained through secure data storage, anonymization, and regulatory compliance with local data protection laws.

The findings from HYIMPACT will provide valuable insights into the long-term real-world effectiveness of Nebilet® in managing hypertension. By analyzing treatment adherence, quality of life, and cardiovascular outcomes over time, this study will contribute to optimizing hypertension treatment strategies and improving patient care across diverse healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age with either newly diagnosed or uncontrolled hypertension (office SBP ≥140 and/or DBP ≥90 mmHg recorded at the time of screening) as per ESC/ESH guidelines 2018.
* Hypertensive patients - with or without cardiovascular comorbidities (such as coronary artery disease, heart failure, peripheral artery disease, cerebrovascular disease, arrhythmias, and valvular heart disease) - who are newly prescribed or are already on Nebilet based treatment (no more than for 2 weeks at screening).
* Hypertensive patients willing to provide consent to participate in the study.
* Women of reproductive age who are willing to use adequate means of contraception.

Exclusion Criteria:

* Patients with recent cardiovascular event within less than 3 months.
* Patient with heart failure based on New York Heart Association (NYHA) Functional Classification- Class IV.
* Patients with contraindications to Nebilet based treatment as per respective Summary of Product Characteristic (SmPC) which in the treating physician's judgment may jeopardize the subject by his or her participation in this study or may hamper his or her ability to perform and complete procedures required in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from South-East Asia countries will be enrolled.
  The names of the participating countries are as follows:
  1. Taiwan
  2. Indonesia
  3. South Korea
  4. Philippines
  5. Thailand
  6. Malaysia
  7. Vietnam
Sampling Method: Non-Probability Sample
Enrollment: 4537 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in mean sitting systolic blood pressure from baseline to one year of treatment in hypertensive patients on Nebilet based treatment. | Baseline to 12 months
  Blood pressure of the study patients will be recorded and documented within a time period of every 3 months since baseline visit.

SECONDARY OUTCOMES:
To assess the impact of Nebilet based treatment in changing diastolic BP (DBP) in hypertensive patients in real-world setting from baseline to one year of treatment. | Baseline to 12 months
  Change in mean sitting Diastolic Blood Pressure (DBP) from baseline to one year of treatment in hypertensive patients on Nebilet based combination treatment.
Change in mean sitting SBP and DBP from baseline to two years and at the end of three years in hypertensive patients on Nebilet based treatment. | Baseline to 24 months and 36 months
  Change in mean sitting SBP and DBP from baseline to 24 months and 36 months of treatment.
To evaluate the proportions of patients achieving target BP goal (<140/90 mm Hg) at different time points (12 months, 24 months, and 36 months of treatment) with Nebilet based as combination treatment. | 12, 24 and 36 months
  For hypertensive patients with coronary artery disease (CAD), the age-wise SBP control goal is ≤130 mmHg in 18-64 years age-group, and 130 -140 mmHg in ≥65 years age group. Whereas the DBP control goal in these patients is 70-79 mmHg for all age groups.
To assess the association of various risk factors (diabetes, obesity, and hypercholesterolemia) on development of major cardiac events in patients who achieve BP control over a period of 36 months. | 36 months
  The number of Major Adverse Cardiac Events (MACE) such as acute myocardial infarction, acute coronary syndrome, stroke, heart failure, all-cause death and cardiovascular death in patients who achieved target BP control over a period of three years by categorizing the patients as per the risk factors (diabetes, obesity, and hypercholesterolemia).
To study the prescription patterns of Nebilet®-based treatment in terms of frequency per day in real-world settings. | 36 months
  Understanding the prescription patterns of Nebilet in the participating South-East Asia countries.
To study the prescription patterns of Nebilet®-based treatment in terms of dose in milligrams in real-world settings. | 36 months
  Understanding the prescription patterns of Nebilet in the participating South-East Asia countries.
To study the prescription patterns or Nebilet®-based treatment in terms of treatment duration in months, in real-world settings. | 36 months
  Understanding the prescription patterns of Nebilet in the participating South-East Asia countries.
To assess the impact of Nebilet®-based treatment on the quality-of-life of patients using MINICHAL questionnaire. | Baseline, 12 months, 24 months and 36 months
  Understanding the prescription patterns of Nebilet in the participating South-East Asia countries.
To assess the patient-reported outcomes using a short form 36 health survey (SF-36 questionnaire) . | Baseline, 12 month, 24 month, and 36 month
  Assessment of patient reported outcome using short from 36 health survey questionnaire.
To assess patient adherence to treatment by an 8-item Morisky Medication Adherence Scale every 3 months after baseline, till 36 months. | 3 month, 6 month, 9 month, 12 month, 15 month, 18 month, 21 month, 24 month, 27 month, 30 month, 33 month, 36 month
  Assessment of patient adherence to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Radhika Mehta, Study Director — A. Menarini Asia-Pacific Holding Pte Ltd
Locations (49):
- Indonesia (15):
  - Telogorejo Hospital, Semarang, Central Java
  - Bethesda Hospital, Yogyakarta, Central Java
  - Panti rapih Hospital, Yogyakarta, Central Java
  - Husada Utama Hospital, Surabaya, East Java
  - Premere Surabaya Hospital, Surabaya, East Java
  - National Cardiovascular Center Harapan Kita Hospital, Jakarta, Jakarta Special Capital Region
  - Metropolitan Medical Centre Hospital, Jakarta, Jakarta Special Capital Region
  - Bidakara Medical Centre, Selatan, Jakarta Special Capital Region
  - PT Ekamas International Hospital, Pekanbaru, Riau
  - Stella Maris Hospital, Makassar, South Sulawasi
  - Bukit Asam Medika Hospital, Palembang, South Sumatra
  - Advent Hospital, Bandung, West Java
  - Borromeus Hospital, Bandung, West Java
  - RSUD Syamsudin Hospital, Sukabumi, West Java
  - Semen Padang Hospital, Padang, West Sumatra
- Malaysia (6):
  - DrThong,Leow,Chiam & Partners, Kuala Lumpur, Kuala Lumpur
  - Klinik Pembangunan Sdn. Bhd, Kuala Lumpur, Kuala Lumpur
  - Pantai HKL, Kuala Lumpur, Kuala Lumpur
  - Columbia Asia Hospital Seremban, Seremban, Negeri Sembilan
  - Mawar Medical Centre, Seremban, Negeri Sembilan
  - Bukit Tinggi Medical Centre, Klang, Selangor
- Philippines (2):
  - Mary Mediatrix Medical Center, Lipa, Batangas
  - Veterans Memorial Medical Center, Quezon City, Manila
- South Korea (3):
  - Kangbuk Samsung Hospital, Seoul, Jongno District Seoul
  - Eunpyeong St. Mary's Hospital, Seoul, Seoul
  - Chonnam National University Hospital, Gwangju
- Taiwan (13):
  - Far Eastern Memorial Hospital (FEMH), New Taipei City, Banqiao
  - Changhua Christian Hospital (CCH), Changhua, Changhua County
  - Chang Gung Memorial Hospital-Chiayi branch (CGMH-CY), Pozi, Chiayi County
  - Chung Gung Memorial Hospital-Linkou Branch (CGMH-LK), Taoyuan District, Guishan District
  - Hualien Tzu-Chi Hospital (HTCH), Hualien City, Hualien County
  - Asia University Hospital (AUH), Taipei, Nangang Dist.
  - National Cheng Kung University Hospital (NCKUH), Tainan, North District
  - Kaohsiung Medical University Hospital (KMUH), Kaohsiung City, Sanmin District
  - Taipei Medical University Hospital (TMUH), Taipei, Xinyi District
  - Taichung Veterans General Hospital (TVGH), Taichung, Xitun District
  - Chi-Mei Medical Center (CMC), Tainan, Yongkang Dist.
  - MacKay Memorial Hospital (MMH), Taipei, Zhongshan District
  - National Taiwan University Hospital (NTUH), Taipei, Zhongzheng District
- Thailand (6):
  - Vajira Hospital Namindradhiraj University, Dusit, Bangkok
  - Wetchakarunrasm Hospital, Nong Chok, Bangkok
  - Burapha University, Chon Buri, Changwat Chon Buri
  - Central Chet Institute, Nonthaburi, Changwat Nonthaburi
  - Chiang Mai University, Chiang Mai, Chiang Mai
  - Anand Mahidhol Hospital, Lopburi, Lopaburi
- Vietnam (4):
  - CanTho General Hospital, Can Tho, Can Tho City
  - Hanoi Heart Hospital, Hanoi, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City, Ho Chi Minh
  - Hue Central Hospital, Huế, Hue

IPD SHARING:
Plan to Share IPD: Undecided